CLINICAL TRIAL: NCT06520566
Title: Holistic Care Partners: A Black Woman-led Nurse Navigation Program to Improve Care, Reduce Harm, and Enhance Perinatal Wellbeing for Black Birthing People
Brief Title: Holistic Care Partner Program Feasibility and Acceptability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-00821; 1R21NR020960-01 (NIH)
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Maternal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Black Birthing Patients enrolled in Holistic Care Partner Program (HCP) (Experimental): Black birthing patients enrolled in HCP will be invited to participate in a brief survey and/or a qualitative interview throughout 1 year of their enrollment.
  Interventions: Behavioral: Holistic care partner perinatal nurse navigation

INTERVENTIONS:
Behavioral: Holistic care partner perinatal nurse navigation — The nurse navigators assess patient medical, social, and structural needs at enrollment, 20-, 28-, and 36-weeks gestation; and at 1-week, and 3, 6, and 9 months postpartum. They provide coordination, support, and referrals, and enhanced communication with or escalate concerns to the primary physician as indicated. The nurse navigator tailors additional visits to the individual needs of the patients (for example, managing comorbidities, social isolation, breastfeeding support). Participants also have access to a Black woman-led support group during pregnancy and the first postpartum year, and access to Black woman-led childbirth and lactation classes.

SUMMARY:
The study aims to build on the knowledge of the United States' ongoing maternal health crisis for Black birthing people. The study team will take a holistic focused approach to build on the experiences of Black women perinatal nurses, Black women/birthing people, and their care partners enrolled in the Holistic Care Partner Program (HCP) to understand the program's feasibility and acceptability. HCP was developed at NYU Langone Health by Blank women-led perinatal nurses to address the effects of obstetric racism and the associated fear of pregnancy and birth faced by Black women and birthing people. Utilizing a mixed-methods approach, the study will focus on understanding HCP's acceptability and feasibility via surveys and qualitative interviews with Black women and birthing people and their partners/support persons to identify strategies and recommendations for intervention improvement. Exploratory analysis of maternal and infant outcomes will be conducted using a propensity score matched historical control group.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as Black or within the Black/African Diaspora
2. Enrolled in the HCP program while pregnant or within 6 weeks postpartum
3. Enrolled in the Faculty Group Practice at NYU Langone Health (NYULH) for obstetric care
4. Plan to give birth at NYULH Tisch or gave birth at NYULH Tisch if postpartum at screening.
5. Comfortable reading and/or speaking English (approximately 95% of Black women speak English)
6. Are 18 years or older

Exclusion Criteria:

1. Does not identify as Black or within the Black/African Diaspora
2. Did not enroll in the HCP program while pregnant or within 6 weeks postpartum.
3. Not enrolled in the FGP NYULH for obstetric care
4. Does not plan to give birth at NYULH Tisch or did not give birth at NYULH Tisch if postpartum at time of screening.
5. Is not 18 years or older
6. Multiple gestation
7. Significant fetal anomaly requiring exceptional care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the study | Visit 4 (9-12 months postpartum)
Theoretical Framework for Acceptability (TFA) questionnaire score | Visit 3 (6-12 weeks postpartum)
  Anticipated and experienced acceptability will be measured using the Theoretical Framework for Acceptability questionnaire. This is a 13-item Likert-type questionnaire designed to assess acceptability of the intervention from the participants' perspective along the 7 component constructs (affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy).
  Total score ranges from 13-65, with higher scores indicating greater acceptability of the intervention.
Attendance rate for nurse navigator visits | Visit 4 (9-12 months postpartum)
Attendance rate at lactation classes | Visit 4 (9-12 months postpartum)
Attendance rate at the support group | Visit 4 (9-12 months postpartum)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Lyndon, PhD, RNC, FAAN, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The redacted interview transcripts from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data and who provide a methodologically sound proposal executes a data use agreement with NYU Langone Health. Requests may be directed to: al6148@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and who provide a methodologically sound proposal will be provided access upon reasonable request. Requests should be directed to al6148@nyu.edu. To gain access, data requestors will need to sign a data access agreement.